CLINICAL TRIAL: NCT01011894
Title: A Phase II Study of Lenalidomide in Patients With Chronic Lymphocytic Leukemia Older Than 65 Years of Age
Brief Title: Lenalidomide in Patients With Chronic Lymphocytic Leukemia Older Than 65 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-045
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia
Keywords: Lenalidomide; CLL; 09-045
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Lenalidomide

ARMS (1):
- pts getting lenalidomide (Experimental): Patients with intermediate or high-risk chronic lymphocytic leukemia (≥ 65 years old) will receive lenalidomide until disease progression at the 20mg dose level (recognizing that progression at this dose requires non-protocol alternate therapy) or unacceptable toxicity.
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Lenalidomide will be administered orally at a starting dose of 2.5mg once daily, days 1-28. Patients will be evaluated prior to treatment and at 4 weeks, 8 weeks, 12 weeks, 16 weeks and at a minimum of 4 weeks thereafter until removal from study. Patients with stable disease or better will continue at their current dose unless they experience toxicity requiring dose reduction. For those patients who have progressive disease on their current dose and have no dose-limiting toxicity, their dose will be increased from 2.5mg, to 5mg, to 10mg, to 15mg, to 20mg one dose level at a time not more frequently than once every 4 weeks. The maximum dose will be 20mg.
  Other Names: Responding patients and those with stable disease will continue lenalidomide; at their current dose level and will continue to be evaluated at the above; time points. Following 16 weeks, evaluation will occur at a minimum of every 4 weeks until; removal from the study. Patients who have stable disease or are responding following the first; year of treatment will be required to have monthly blood work but can be seen at no less than 3; month intervals.

SUMMARY:
The purpose of this study is to:

Determine the likelihood that lenalidomide will adequately control the disease for at least one year.

Lenalidomide is a drug that alters the immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. Lenalidomide is approved by the Food and Drug Administration (FDA) for the treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for patients with multiple myeloma (MM) who have received at least 1 prior therapy. MDS and MM are cancers of the blood. It is currently being tested in a variety of cancer conditions.

In this case it is considered experimental. The lenalidomide being administered in this study is not a commercially marketed product. Although it is expected to be very similar in safety and activity to the commercially marketed drug, it is possible that some differences may exist. Because this is not a commercially marketed drug, lenalidomide can only be administered to patients enrolled in this clinical trial and may only be administered under the direction of physicians who are investigators in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either previously untreated or treated disease must have either intermediate or high-risk chronic lymphocytic leukemia as defined by the three-stage Rai system. Patients with Rai intermediate risk disease should meet the criteria for active disease as outlined by the NCI Working Group guidelines (including weight loss, fatigue, fevers, evidence of progressive marrow failure, splenomegaly, progressive lymphadenopathy, or progressive lymphocytosis with a rapid doubling time)(49).
* MSKCC pathologist must confirm patient's disease.
* To be considered CLL the patient must have an absolute lymphocytosis in the blood of at least 5,000 lymphocytes per microliter, or bone marrow lymphocytosis greater than or equal to 30% of all nucleated cells
* Immunophenotypic (or immunohistochemical) analysis of the malignant lymphocytes should demonstrate that the cells are B-cells. Typically these cells should also express CD5 and CD23. It is recognized that an occasional patient with CLL may have a slightly aberrant immunophenotype. All such cases need to be reviewed with the principal investigator prior to being registered for the study. Patients with small lymphocytic lymphoma (CLL type) will be eligible for this study.
* Age ≥ 65 years of age.
* Karnofsky performance status ≥ 50%
* ANC ≥ 0.8 and platelet count ≥ 30,000
* Total creatinine ≤ 2.0mg/dl or creatinine clearance ≥ 30ml/min.
* Total bilirubin ≤ 3.0 mg/dL (not attributable to autoimmune hemolytic anemia).
* Signed informed consent, which indicates the investigational nature of this study, is required.
* No patient may be entered onto the study without consultation with the principal investigator or his designee.
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.

Exclusion Criteria:

* Patients with significant active infections.
* Men should use effective contraception.
* Patients known positive for HIV or with active infection from hepatitis, A, B, or C.
* Concomitant chemotherapy or radiotherapy while on protocol.
* Evidence of laboratory TLS by Cairo-Bishop Definition of Tumor Lysis Syndrome.
* History of thromboembolic disease within the past 6 months, regardless of anti-coagulation.
* Myocardial infarction within 6 months prior to enrollment, or New York Hospital Association (NYHA) Class III or IV heart failure , uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11-06; Primary Completion 2016-02-23 (Actual); Study Completion 2016-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renier Brentjens, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 11/6/2009, Protocol Closed to Accrual 2/26/2013, Primary Completion Date 2/23/2016, Recruitment location is the medical clinic
Groups:
- Intermediate or High Risk Chronic Lymphocytic Leukemia: This is a single-arm open label study designed to assess the efficacy of continuous lenalidomide therapy in patient >/= 65 years old.
Period: Overall Study
Arm/Group | Intermediate or High Risk Chronic Lymphocytic Leukemia
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intermediate or High Risk Chronic Lymphocytic Leukemia
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Response
Description: The major criteria for determination of response to therapy in patients with CLL include physical examination and examination of the peripheral blood and bone marrow. Complete Response (CR): Absence of lymphadenopathy, hepatomegaly or splenomegaly by physical examination and appropriate radiographic techniques (if abnormal pre-treatment), No constitutional symptoms, ANC >/= 1,500/ul, platelets> 100,000/ul, Hgb>11gm/dl (untransfused); Partial Response (PR): >50% decrease in peripheral blood lymphocyte count from the pre-treatment baseline value, reduction in lymphadenopathy, reduction in size of the liver and/or the spleen; Progressive Disease (PD): Characterized by at least one of the following: > 50% increase in the sum of the products of at least 2 lymph nodes on at least 2 consecutive exams at least 2 weeks apart. At least 1 node must be >/= to 2cm in size, Appearance of new palpable LN, > 50% increase in size of liver or spleen determined by measurement below the respective costal
Time Frame: 2 years
Population: 20 participants had Stable Disease, 3 had Progression of Disease, 3 were not evaluable due to toxicity
Measure: Count of Participants; unit: Participants
Groups:
- Participants Receiving Lenalidomide: Patients with intermediate or high-risk chronic lymphocytic leukemia (≥ 65 years old) will receive lenalidomide until disease progression at the 20mg dose level (recognizing that progression at this dose requires non-protocol alternate therapy) or unacceptable toxicity.
Arm/Group | Participants Receiving Lenalidomide
Number analyzed (Participants) | 26
Participants
  Stable Disease | 20
  Progressive Disease | 3
  Not Evaluable | 3

ADVERSE EVENTS:
Arm/Group | Intermediate or High Risk Chronic Lymphocytic Leukemia
Serious Adverse Events (participants affected / at risk) | 11/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intermediate or High Risk Chronic Lymphocytic Leukemia (N=26)
ALT, SGPT (Blood and lymphatic system disorders) | 1
Creatinine increased (Metabolism and nutrition disorders) | 1
Dizziness (General disorders) | 1
Fatigue (General disorders) | 3
Febrile neutropenia (General disorders) | 1
Headache (General disorders) | 1
Skin infection (Skin and subcutaneous tissue disorders) | 1
Pneumonia (General disorders) | 4
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3
Platelet count decreased (Blood and lymphatic system disorders) | 1
Thrombosis/thrombus/embolism (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intermediate or High Risk Chronic Lymphocytic Leukemia (N=26)
Neutrophil count decreased (Investigations) | 19
Platelet count decreased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 4
Anemia (Blood and lymphatic system disorders) | 3
Alanine aminotransferase increased (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
INR increased (Investigations) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes